CLINICAL TRIAL: NCT00540592
Title: Observer Blind Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' Influenza Vaccine GSK576389A With Various Formulations in Adults Aged 65 Years and Above
Brief Title: Immunogenicity and Safety Study to Evaluate Different Formulations of GSK Biologicals' Influenza Vaccine GSK576389A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110847
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza vaccine GSK576389A; Influenza infection; Fluarix
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (10):
- Influenza vaccine GSK576389A formulation 1 Group (Experimental): Subjects aged ≥65 years received one dose of formulation 1 of the adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A
- Influenza vaccine GSK576389A formulation 2 Group (Experimental): Subjects aged ≥65 years received one dose of formulation 2 of the adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A
- Influenza vaccine GSK576389A formulation 3 Group (Experimental): Subjects aged ≥65 years received one dose of formulation 3 of the adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A
- Influenza vaccine GSK576389A formulation 4 Group (Experimental): Subjects aged ≥65 years received one dose of formulation 4 of the adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A
- Influenza vaccine GSK576389A formulation 5 Group (Experimental): Subjects aged ≥65 years received one dose of formulation 5 of the adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A
- Influenza vaccine GSK576389A formulation 6 Group (Experimental): Subjects aged ≥65 years received one dose of formulation 6 of the adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A
- Influenza vaccine GSK576389A formulation 7 Group (Experimental): Subjects aged ≥65 years received one dose of formulation 7 of the adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A
- Influenza vaccine GSK576389A formulation 8 Group (Experimental): Subjects aged ≥65 years received one dose of formulation 8 of the adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A
- Fluarix elderly Group (Active Comparator): Subjects aged ≥65 years received one dose of Fluarix vaccine.
  Interventions: Biological: Fluarix
- Fluarix young Group (Active Comparator): Subjects aged 18-40 years received one dose of Fluarix vaccine.
  Interventions: Biological: Fluarix

INTERVENTIONS:
Biological: GlaxoSmithKline Biologicals' influenza vaccine GSK576389A — Single dose, Intramuscular injection, 8 different formulations were tested (one per group)
  Arms: Influenza vaccine GSK576389A formulation 1 Group; Influenza vaccine GSK576389A formulation 2 Group; Influenza vaccine GSK576389A formulation 3 Group; Influenza vaccine GSK576389A formulation 4 Group; Influenza vaccine GSK576389A formulation 5 Group; Influenza vaccine GSK576389A formulation 6 Group; Influenza vaccine GSK576389A formulation 7 Group; Influenza vaccine GSK576389A formulation 8 Group
Biological: Fluarix — Single dose, Intramuscular injection
  Arms: Fluarix elderly Group; Fluarix young Group

SUMMARY:
In order to find the formulation leading to a maximal increase of the immune response while maintaining an acceptable safety profile, this study is designed to evaluate the immunogenicity, safety and reactogenicity of the different formulations of GSK Biologicals' influenza vaccine administered in adults aged 65 years and older compared to Fluarix.

DETAILED DESCRIPTION:
There are 10 parallel groups: 9 observer blinded groups with subjects 65 years and older receiving an investigational vaccine or Fluarix, and 1 open group with subjects between 18 and 40 years old receiving Fluarix. CMI response will be determined for a subset only.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 18-40 years old or 65 years or older at the time of the vaccination.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical evaluation (medical history and medical history directed examination) before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to vaccination, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study.
* Planned administration of a vaccine not foreseen by the study protocol during the entire study period.
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period.
* Vaccination against influenza since January 2007 (with 2007/2008 or 2006/2007 influenza vaccine).
* Administration of more than 14 days of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Hypersensitivity to a previous dose of influenza vaccine.
* Allergy to any component of the vaccine.
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality.
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e. axillary temperature<37.5ºC (99.5ºF).
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the study vaccine or planned administration during the study.
* Any medical conditions in which IM injections are contraindicated.
* Lactating female or female planning to become pregnant or to discontinue contraceptive precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2007 (Actual)
Dates: Start 2007-10-08; Primary Completion 2008-06-10 (Actual); Study Completion 2008-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- Germany (16):
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Rudersberg, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Rotterdam, Netherlands
- Sweden (3):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Uppsala
- United Kingdom (5):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Clydebank, Glasgow
  - GSK Investigational Site, Edgbaston, Birmingham
  - GSK Investigational Site, Waterloo, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Rumke HC, Richardus JH, Rombo L, Pauksens K, Plassmann G, Durand C, Devaster JM, Dewe W, Oostvogels L. Selection of an adjuvant for seasonal influenza vaccine in elderly people: modelling immunogenicity from a randomized trial. BMC Infect Dis. 2013 Jul 26;13:348. doi: 10.1186/1471-2334-13-348. PMID 23890405
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 110847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110847 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Started | 204 | 202 | 202 | 202 | 199 | 198 | 198 | 199 | 200 | 203
Completed at Day 180 | 200 | 201 | 197 | 197 | 195 | 198 | 196 | 193 | 198 | 189
Completed | 202 | 201 | 201 | 201 | 198 | 198 | 198 | 198 | 199 | 201
Not Completed | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group | Total
Number analyzed (Participants) | 204 | 202 | 202 | 202 | 199 | 198 | 198 | 199 | 200 | 203 | 2007
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.7 (5.75) | 72.6 (5.16) | 72.4 (5.62) | 72.9 (6.09) | 72.6 (5.66) | 72.7 (5.56) | 72.6 (5.67) | 73.0 (6.03) | 72.7 (5.43) | 27.4 (6.25) | 68.11 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 109 | 105 | 100 | 89 | 102 | 96 | 95 | 90 | 103 | 984
  Male | 109 | 93 | 97 | 102 | 110 | 96 | 102 | 104 | 110 | 100 | 1023

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers
Description: Antibody titers were expressed as Geometric mean titers (GMTs) against each of the 3 vaccine strains in greater than or equal to 65 years age groups only. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 21
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity HI which included all evaluable subjects for whom data concerning immunogenicity HI outcome measures were available at day 21.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 191 | 192 | 189 | 194 | 192 | 193 | 192 | 189 | 188 | 0
titer
  A/Solomon Islands strain | 82.3 [69.7 to 97.1] | 102.2 [87.0 to 119.9] | 98.2 [84.3 to 114.3] | 91.7 [76.9 to 109.3] | 113.2 [96.0 to 133.6] | 114.4 [97.1 to 134.8] | 78.5 [65.9 to 93.5] | 111.8 [93.3 to 134.0] | 59.6 [49.6 to 71.7] |
  A/Wisconsin strain | 276.2 [238.8 to 319.6] | 350.2 [298.0 to 411.4] | 351.3 [304.8 to 404.8] | 309.2 [264.9 to 361.0] | 331.1 [289.6 to 378.6] | 438.1 [379.7 to 505.4] | 263.3 [225.3 to 307.7] | 347.5 [296.4 to 407.3] | 186.7 [158.0 to 220.7] |
  B/Malaysia strain | 147.1 [129.1 to 167.6] | 163.1 [142.5 to 186.6] | 172.1 [149.9 to 197.6] | 152.4 [134.4 to 172.7] | 181.4 [158.9 to 207.1] | 202.0 [179.7 to 227.1] | 155.7 [134.8 to 179.8] | 174.6 [152.0 to 200.7] | 153.0 [135.2 to 173.1] |

2. Secondary Outcome: HI Antibody Titers at Day 0 and Day 21
Description: Antibody titers were expressed as GMTs in all the vaccine groups. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 191 | 192 | 189 | 194 | 192 | 193 | 192 | 189 | 188 | 197
titer
  A/Solomon Islands strain at Day 0 | 10.6 [9.3 to 12.2] | 10.8 [9.4 to 12.4] | 10.1 [8.8 to 11.5] | 10.6 [9.3 to 12.1] | 12.0 [10.3 to 14.0] | 9.9 [8.6 to 11.3] | 10.2 [8.9 to 11.7] | 10.3 [9.0 to 11.9] | 10.7 [9.2 to 12.4] | 21.3 [17.1 to 26.5]
  A/Solomon Islands strain at Day 21 | 82.3 [69.7 to 97.1] | 102.2 [87.0 to 119.9] | 98.2 [84.3 to 114.3] | 91.7 [76.9 to 109.3] | 113.2 [96.0 to 133.6] | 114.4 [97.1 to 134.8] | 78.5 [65.9 to 93.5] | 111.8 [93.3 to 134.0] | 59.6 [49.6 to 71.7] | 271.6 [224.6 to 328.4]
  A/Wisconsin strain at Day 0 | 59.9 [49.5 to 72.4] | 51.2 [41.9 to 62.4] | 44.4 [36.5 to 54.0] | 65.7 [53.7 to 80.4] | 61.1 [50.6 to 73.8] | 55.8 [46.2 to 67.4] | 54.6 [44.5 to 67.0] | 57.8 [47.1 to 70.9] | 61.0 [49.8 to 74.7] | 47.8 [39.2 to 58.4]
  A/Wisconsin strain at Day 21 | 276.2 [238.8 to 319.6] | 350.2 [298.0 to 411.4] | 351.3 [304.8 to 404.8] | 309.2 [264.9 to 361.0] | 331.1 [289.6 to 378.6] | 438.1 [379.7 to 505.4] | 263.3 [225.3 to 307.7] | 347.5 [296.4 to 407.3] | 186.7 [158.0 to 220.7] | 380.2 [331.6 to 435.9]
  B/Malaysia strain at Day 0 | 58.6 [49.8 to 68.9] | 53.7 [45.7 to 63.2] | 57.0 [48.2 to 67.5] | 62.6 [53.3 to 73.4] | 77.8 [66.0 to 91.7] | 62.9 [53.9 to 73.4] | 58.2 [49.0 to 69.1] | 62.6 [53.0 to 74.0] | 66.5 [56.5 to 78.3] | 23.4 [19.1 to 28.7]
  B/Malaysia strain at Day 21 | 147.1 [129.1 to 167.6] | 163.1 [142.5 to 186.6] | 172.1 [149.9 to 197.6] | 152.4 [134.4 to 172.7] | 181.4 [158.9 to 207.1] | 202.0 [179.7 to 227.1] | 155.7 [134.8 to 179.8] | 174.6 [152.0 to 200.7] | 153.0 [135.2 to 173.1] | 281.9 [241.7 to 328.7]

3. Secondary Outcome: HI Antibody Titers at Day 180
Description: as for outcome 2
Time Frame: At Day 180
Population: Analysis was performed on According-to-Protocol (ATP) cohort for persistence for HI which included all evaluable subjects for whom data concerning immunogenicity HI outcome measures were available at day 180.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 186 | 186 | 180 | 184 | 180 | 187 | 187 | 174 | 181 | 165
titer
  A/Solomon Islands strain | 30.6 [25.8 to 36.3] | 35.1 [29.7 to 41.5] | 36.3 [30.7 to 42.8] | 32.5 [27.6 to 38.2] | 40.4 [34.1 to 47.9] | 33.7 [28.6 to 39.7] | 29.9 [25.5 to 35.0] | 39.8 [33.6 to 47.2] | 23.7 [20.3 to 27.7] | 114.7 [91.8 to 143.5]
  A/Wisconsin strain | 131.5 [112.6 to 153.5] | 139.8 [118.1 to 165.5] | 133.4 [112.7 to 158.1] | 134.0 [113.1 to 158.7] | 144.7 [124.9 to 167.5] | 181.4 [156.5 to 210.3] | 118.2 [99.8 to 140.0] | 145.3 [121.9 to 173.2] | 92.5 [78.7 to 108.6] | 193.2 [163.5 to 228.3]
  B/Malaysia strain | 92.7 [81.2 to 106.0] | 94.3 [81.6 to 109.1] | 100.9 [87.7 to 116.1] | 87.4 [75.9 to 100.6] | 109.2 [94.9 to 125.6] | 111.4 [97.2 to 127.6] | 89.0 [76.1 to 104.0] | 97.7 [84.7 to 112.7] | 96.6 [83.8 to 111.3] | 132.4 [110.2 to 159.0]

4. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies at Day 21
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 191 | 191 | 189 | 194 | 192 | 193 | 192 | 189 | 187 | 197
Subjects
  A/Solomon Islands strain | 133 | 138 | 154 | 130 | 142 | 151 | 129 | 146 | 99 | 135
  A/Wisconsin strain | 108 | 124 | 141 | 104 | 124 | 142 | 110 | 131 | 69 | 130
  B/Malaysia strain | 47 | 73 | 65 | 44 | 45 | 79 | 50 | 55 | 47 | 147

5. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies at Day 180
Description: as for outcome 4
Time Frame: At Day 180
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 186 | 186 | 180 | 184 | 180 | 187 | 187 | 174 | 180 | 165
Subjects
  A/Solomon Islands strain | 64 | 73 | 74 | 68 | 60 | 77 | 60 | 67 | 42 | 90
  A/Wisconsin strain | 47 | 59 | 61 | 46 | 50 | 74 | 37 | 49 | 23 | 74
  B/Malaysia strain | 23 | 23 | 25 | 19 | 16 | 32 | 19 | 20 | 17 | 90

6. Secondary Outcome: HI Antibody Seroconversion Factors at Day 21
Description: Seroconversion factors were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 191 | 191 | 189 | 194 | 192 | 193 | 192 | 189 | 187 | 197
fold increase
  A/Solomon Islands strain | 7.7 [6.5 to 9.2] | 9.4 [7.8 to 11.3] | 9.8 [8.3 to 11.5] | 8.6 [7.2 to 10.4] | 9.4 [8.0 to 11.1] | 11.6 [9.7 to 13.9] | 7.7 [6.5 to 9.2] | 10.8 [9.0 to 13.0] | 5.6 [4.7 to 6.8] | 12.8 [10.0 to 16.3]
  A/Wisconsin strain | 4.6 [3.9 to 5.4] | 6.8 [5.6 to 8.1] | 7.9 [6.6 to 9.5] | 4.7 [4.0 to 5.5] | 5.4 [4.6 to 6.3] | 7.8 [6.5 to 9.5] | 4.8 [4.1 to 5.7] | 6.0 [5.1 to 7.1] | 3.1 [2.6 to 3.6] | 7.9 [6.4 to 9.8]
  B/Malaysia strain | 2.5 [2.2 to 2.8] | 3.0 [2.6 to 3.5] | 3.0 [2.6 to 3.5] | 2.4 [2.2 to 2.8] | 2.3 [2.1 to 2.6] | 3.2 [2.8 to 3.7] | 2.7 [2.3 to 3.1] | 2.8 [2.4 to 3.2] | 2.3 [2.0 to 2.6] | 12.0 [9.7 to 15.0]

7. Secondary Outcome: HI Antibody Seroconversion Factors at Day 180
Description: as for outcome 6
Time Frame: At Day 180
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 186 | 186 | 180 | 184 | 180 | 187 | 187 | 174 | 180 | 165
fold increase
  A/Solomon Islands strain | 2.9 [2.5 to 3.4] | 3.3 [2.8 to 3.9] | 3.5 [3.1 to 4.1] | 3.0 [2.6 to 3.5] | 3.3 [2.9 to 3.8] | 3.5 [2.9 to 4.1] | 2.9 [2.5 to 3.3] | 3.8 [3.2 to 4.4] | 2.2 [1.9 to 2.6] | 5.7 [4.5 to 7.2]
  A/Wisconsin strain | 2.2 [1.9 to 2.6] | 2.7 [2.3 to 3.1] | 2.9 [2.5 to 3.3] | 2.0 [1.8 to 2.3] | 2.4 [2.1 to 2.7] | 3.1 [2.7 to 3.6] | 2.1 [1.8 to 2.4] | 2.5 [2.2 to 2.9] | 1.6 [1.4 to 1.8] | 4.0 [3.2 to 5.0]
  B/Malaysia strain | 1.7 [1.5 to 1.9] | 1.7 [1.5 to 1.9] | 1.7 [1.5 to 1.9] | 1.4 [1.3 to 1.6] | 1.4 [1.3 to 1.6] | 1.8 [1.6 to 2.0] | 1.5 [1.4 to 1.7] | 1.6 [1.4 to 1.8] | 1.5 [1.3 to 1.7] | 5.6 [4.5 to 7.0]

8. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies at Day 0 and 21
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 191 | 192 | 189 | 194 | 192 | 193 | 192 | 189 | 188 | 197
Subjects
  A/Solomon Islands strain at Day 0 | 27 | 31 | 25 | 33 | 44 | 23 | 22 | 26 | 31 | 69
  A/Solomon Islands strain at Day 21 | 160 | 168 | 171 | 158 | 169 | 172 | 153 | 163 | 132 | 182
  A/Wisconsin strain at Day 0 | 133 | 124 | 113 | 139 | 131 | 139 | 130 | 134 | 132 | 122
  A/Wisconsin strain at Day 21 | 188 | 189 | 188 | 190 | 192 | 191 | 187 | 185 | 179 | 197
  B/Malaysia strain at Day 0 | 138 | 140 | 138 | 148 | 156 | 149 | 139 | 145 | 144 | 77
  B/Malaysia strain at Day 21 | 183 | 183 | 184 | 187 | 186 | 192 | 182 | 184 | 183 | 195

9. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies at Day 180
Description: as for outcome 8
Time Frame: At Day 180
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 186 | 186 | 180 | 184 | 180 | 187 | 187 | 174 | 181 | 165
Subjects
  A/Solomon Islands strain | 94 | 111 | 105 | 105 | 103 | 104 | 100 | 100 | 77 | 135
  A/Wisconsin strain | 172 | 170 | 162 | 164 | 170 | 179 | 166 | 160 | 156 | 158
  B/Malaysia strain | 167 | 166 | 168 | 168 | 166 | 176 | 158 | 162 | 162 | 144

10. Secondary Outcome: The Geometric Mean (GM) Number of Influenza-specific CD4 T-cells Per Million CD4+ T-cells for Each Vaccine Strain Producing at Least Two Different Immune Markers or Producing Each of the Immune Markers Plus Another Immune Marker at Days 0 and 21
Description: The markers assessed were Cluster of Differentiation 4-All doubles i.e. CD4-All doubles, CD4-CD40Ligand(L), CD4-interferon gamma (CD4-IFNγ), CD4-interleukin 2 (CD4-IL2) and CD4-tumor necrosis factor alpha (CD4-TNFα). The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Days 0 and 21
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity cell mediated immunity (CMI) which included subjects for whom data concerning immunogenicity CMI outcome measures were available at day 21.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD4 T-cells
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 24 | 19 | 25 | 24 | 24 | 23 | 23 | 23 | 23 | 23
cells per million CD4 T-cells
  A/Solomon Islands [CD4-All doubles] at Day 0 | 177.48 (278.18) | 283.18 (319.74) | 204.49 (236.05) | 200.21 (480.41) | 193.35 (324.34) | 177.44 (297.52) | 199.80 (310.58) | 222.58 (282.91) | 156.21 (518.89) | 538.72 (442.78)
  A/Solomon Islands [CD4-All doubles] at Day 21 | 441.16 (517.73) | 856.00 (685.35) | 704.14 (778.07) | 494.63 (883.53) | 483.24 (481.37) | 808.90 (858.38) | 655.32 (616.75) | 797.68 (5271.86) | 536.24 (578.48) | 1027.23 (838.01)
  A/Wisconsin [CD4-All doubles] at Day 0 | 583.77 (563.98) | 488.70 (540.66) | 584.25 (626.26) | 309.67 (517.11) | 538.87 (691.59) | 702.79 (3741.48) | 457.98 (321.69) | 594.26 (598.83) | 427.71 (745.78) | 821.78 (646.48)
  A/Wisconsin [CD4-All doubles] at Day 21 | 1016.63 (990.97) | 1491.86 (899.50) | 1140.56 (955.61) | 1015.18 (1044.87) | 1051.06 (1024.97) | 1998.33 (2730.32) | 1234.37 (830.47) | 1302.34 (3490.03) | 922.62 (1170.30) | 1455.68 (870.69)
  B/Malaysia [CD4-All doubles] at Day 0 | 407.18 (456.82) | 596.53 (400.24) | 500.81 (734.64) | 250.48 (375.23) | 490.56 (546.12) | 259.15 (278.35) | 403.06 (482.16) | 442.39 (315.27) | 301.23 (584.68) | 1098.75 (909.18)
  B/Malaysia [CD4-All doubles] at Day 21 | 1025.01 (736.55) | 1614.14 (953.74) | 1005.72 (1314.69) | 817.57 (675.70) | 1019.48 (698.91) | 1255.53 (941.27) | 1153.76 (699.26) | 1057.60 (4968.52) | 781.66 (880.46) | 1707.62 (1591.31)
  A/Solomon Islands [CD4-CD40L] at Day 0 | 187.19 (277.14) | 285.19 (319.80) | 193.56 (236.01) | 141.26 (500.24) | 192.02 (314.38) | 167.87 (296.47) | 153.91 (311.96) | 165.48 (281.57) | 150.60 (512.37) | 504.55 (441.35)
  A/Solomon Islands [CD4-CD40L] at Day 21 | 418.24 (523.39) | 657.41 (684.48) | 641.98 (752.95) | 471.56 (881.73) | 391.29 (474.16) | 510.16 (871.38) | 599.32 (592.08) | 697.39 (5282.26) | 406.14 (571.70) | 967.83 (848.55)
  A/Wisconsin [CD4-CD40L] at Day 0 | 555.20 (555.43) | 477.12 (531.36) | 527.80 (613.23) | 284.63 (522.58) | 511.21 (679.89) | 587.17 (1872.24) | 418.98 (333.83) | 568.96 (559.46) | 322.37 (713.98) | 742.80 (659.21)
  A/Wisconsin [CD4-CD40L] at Day 21 | 941.04 (994.45) | 1438.93 (881.80) | 1014.97 (933.09) | 940.53 (1065.84) | 977.44 (970.75) | 1763.75 (1858.49) | 1162.09 (715.63) | 1156.07 (3501.25) | 798.75 (1155.23) | 1383.25 (871.98)
  B/Malaysia [CD4-CD40L] at Day 0 | 387.03 (429.86) | 587.72 (396.47) | 446.80 (736.88) | 219.83 (386.13) | 479.21 (550.01) | 256.73 (280.28) | 383.93 (466.87) | 431.32 (319.06) | 342.65 (589.08) | 1076.46 (903.85)
  B/Malaysia [CD4-CD40L] at Day 21 | 926.13 (749.19) | 1570.30 (962.36) | 958.63 (1315.41) | 754.45 (694.91) | 975.92 (710.25) | 1160.31 (959.34) | 1039.13 (699.33) | 957.22 (5023.06) | 707.72 (874.64) | 1614.08 (1617.78)
  A/Solomon Islands [CD4-IFNγ] at Day 0 | 202.65 (195.65) | 190.19 (245.89) | 158.04 (192.23) | 235.01 (355.44) | 171.07 (194.84) | 137.02 (189.76) | 203.95 (254.48) | 184.52 (211.26) | 198.86 (422.78) | 380.34 (384.07)
  A/Solomon Islands [CD4-IFNγ] at Day 21 | 398.57 (370.41) | 636.42 (570.57) | 532.84 (488.63) | 426.15 (660.07) | 379.49 (361.80) | 543.09 (681.65) | 467.66 (450.93) | 576.14 (4664.15) | 442.66 (449.36) | 755.12 (645.89)
  A/Wisconsin [CD4-IFNγ] at Day 0 | 361.99 (378.72) | 350.04 (325.28) | 332.39 (326.71) | 295.56 (424.20) | 243.93 (321.57) | 495.18 (3550.69) | 305.13 (248.40) | 310.45 (276.10) | 272.34 (453.35) | 589.57 (493.89)
  A/Wisconsin [CD4-IFNγ] at Day 21 | 644.07 (707.63) | 891.98 (719.87) | 809.46 (590.21) | 606.43 (745.80) | 651.21 (651.51) | 1293.10 (2390.91) | 718.87 (619.16) | 691.57 (2944.57) | 548.91 (732.46) | 976.96 (643.43)
  B/Malaysia [CD4-IFNγ] at Day 0 | 336.70 (352.20) | 403.08 (319.99) | 322.07 (631.98) | 302.23 (249.59) | 248.66 (236.24) | 237.57 (200.43) | 277.94 (372.05) | 210.23 (266.19) | 256.03 (440.55) | 874.82 (729.66)
  B/Malaysia [CD4-IFNγ] at Day 21 | 716.86 (601.16) | 1163.80 (865.47) | 855.95 (1073.89) | 509.84 (520.06) | 611.65 (527.80) | 852.80 (715.28) | 745.46 (575.21) | 709.84 (4385.83) | 523.15 (697.47) | 1306.18 (1346.37)
  A/Solomon Islands [CD4-IL2] at Day 0 | 181.54 (242.60) | 193.42 (297.22) | 188.29 (215.39) | 150.59 (407.63) | 152.22 (284.11) | 157.54 (255.06) | 161.81 (293.16) | 170.79 (253.02) | 122.12 (451.59) | 356.84 (313.43)
  A/Solomon Islands [CD4-IL2] at Day 21 | 299.14 (421.84) | 664.46 (582.79) | 559.98 (642.32) | 415.13 (691.39) | 409.73 (365.35) | 677.81 (689.59) | 529.19 (520.65) | 678.22 (4760.15) | 461.05 (498.00) | 813.73 (693.31)
  A/Wisconsin [CD4-IL2] at Day 0 | 406.48 (508.99) | 382.61 (428.51) | 516.80 (421.85) | 251.35 (445.04) | 388.89 (560.47) | 532.86 (708.29) | 393.79 (295.93) | 470.64 (443.13) | 343.41 (607.93) | 589.89 (469.14)
  A/Wisconsin [CD4-IL2] at Day 21 | 747.93 (778.49) | 1082.78 (712.53) | 1010.24 (772.39) | 762.07 (766.05) | 792.75 (828.41) | 1425.03 (1236.35) | 908.72 (680.48) | 1041.76 (2883.12) | 733.36 (900.95) | 1061.62 (635.42)
  B/Malaysia [CD4-IL2] at Day 0 | 277.98 (394.46) | 491.65 (369.85) | 434.78 (621.10) | 190.27 (322.46) | 411.11 (457.99) | 269.03 (243.51) | 360.78 (420.71) | 333.95 (309.81) | 221.19 (537.35) | 871.60 (724.64)
  B/Malaysia [CD4-IL2] at Day 21 | 791.31 (616.06) | 1295.22 (856.91) | 992.50 (1134.21) | 692.82 (570.55) | 876.95 (569.97) | 1038.01 (765.73) | 949.33 (588.11) | 872.00 (4655.93) | 695.83 (757.57) | 1348.21 (1359.92)
  A/Solomon Islands [CD4-TNFα] at Day 0 | 91.32 (201.60) | 155.22 (184.44) | 130.19 (152.33) | 124.70 (306.20) | 143.44 (199.20) | 112.41 (169.39) | 100.38 (185.42) | 111.07 (179.39) | 104.10 (311.25) | 234.98 (234.23)
  A/Solomon Islands [CD4-TNFα] at Day 21 | 234.99 (298.31) | 440.26 (451.77) | 333.95 (487.76) | 279.64 (553.81) | 296.79 (289.33) | 336.45 (541.95) | 325.65 (410.44) | 449.86 (3979.03) | 273.66 (355.95) | 490.23 (532.90)
  A/Wisconsin [CD4-TNFα] at Day 0 | 351.26 (450.82) | 458.02 (373.43) | 432.24 (487.63) | 342.30 (455.39) | 404.64 (410.30) | 600.83 (3581.08) | 303.13 (263.25) | 420.75 (422.38) | 327.09 (552.26) | 667.60 (450.65)
  A/Wisconsin [CD4-TNFα] at Day 21 | 712.96 (700.26) | 944.29 (589.91) | 852.44 (637.30) | 623.21 (728.42) | 702.41 (635.67) | 1293.59 (2431.45) | 802.15 (591.12) | 884.71 (2654.95) | 575.97 (723.76) | 995.86 (630.33)
  B/Malaysia [CD4-TNFα] at Day 0 | 203.89 (281.14) | 239.73 (260.28) | 225.66 (501.91) | 118.04 (257.63) | 241.23 (332.43) | 117.51 (175.00) | 152.19 (297.33) | 193.88 (141.46) | 126.64 (402.92) | 605.04 (641.27)
  B/Malaysia [CD4-TNFα] at Day 21 | 509.26 (451.20) | 806.86 (561.77) | 601.64 (763.90) | 312.72 (391.89) | 518.35 (419.60) | 580.98 (579.68) | 547.64 (464.44) | 540.54 (3022.19) | 285.50 (526.85) | 805.41 (1133.76)

11. Secondary Outcome: The GM Number of Influenza-specific CD4 T-cells Per Million CD4+ T-cells for Each Vaccine Strain Producing at Least Two Different Immune Markers or Producing Each of the Immune Markers Plus Another Immune Marker at Day 180
Description: The markers assessed were CD4-All doubles, CD4-CD40L, CD4-IFNγ, CD4-IL2 and CD4-TNFα. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 180
Population: Analysis was performed on According-to-Protocol (ATP) cohort for persistence for cell mediated immunity (CMI) which included subjects for whom data concerning immunogenicity CMI outcome measures were available at day 180.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD4 T-cells
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 21 | 18 | 20 | 17 | 21 | 21 | 19 | 16 | 16 | 19
cells per million CD4 T-cells
  A/Solomon Islands [CD4-All doubles] | 393.50 (359.42) | 348.12 (422.44) | 666.01 (663.86) | 394.45 (508.40) | 432.70 (374.70) | 421.08 (613.81) | 357.66 (470.53) | 224.47 (332.47) | 714.85 (658.37) | 1070.14 (874.71)
  A/Wisconsin [CD4-All doubles] | 802.04 (391.96) | 603.15 (559.07) | 720.91 (829.77) | 463.85 (832.67) | 728.09 (640.63) | 676.69 (785.39) | 670.60 (881.04) | 566.79 (522.16) | 638.11 (929.43) | 1366.02 (966.33)
  B/Malaysia [CD4-All doubles] | 679.05 (4150.67) | 807.74 (629.48) | 807.96 (901.44) | 416.48 (442.15) | 774.07 (452.40) | 423.03 (839.74) | 582.68 (429.62) | 588.22 (334.48) | 742.01 (481.80) | 1304.54 (1096.30)
  A/Solomon Islands [CD4-CD40L] | 348.06 (342.53) | 319.80 (403.11) | 622.84 (626.39) | 361.05 (490.66) | 425.72 (346.49) | 471.70 (566.40) | 353.82 (432.84) | 234.90 (304.83) | 690.69 (642.61) | 999.02 (831.24)
  A/Wisconsin [CD4-CD40L] | 733.96 (397.17) | 576.04 (543.29) | 682.43 (823.68) | 439.97 (825.94) | 680.00 (607.45) | 683.28 (761.14) | 623.11 (800.89) | 554.83 (502.42) | 625.97 (924.73) | 1268.21 (889.54)
  B/Malaysia [CD4-CD40L] | 621.50 (3427.50) | 764.21 (613.38) | 779.35 (887.41) | 394.05 (415.93) | 743.85 (425.01) | 414.76 (732.26) | 592.52 (424.79) | 537.41 (351.86) | 679.16 (486.34) | 1260.62 (1067.54)
  A/Solomon Islands [CD4-IFNγ] | 244.53 (325.64) | 375.03 (308.38) | 392.18 (500.72) | 280.73 (402.63) | 261.43 (263.15) | 338.11 (488.06) | 271.38 (373.04) | 136.97 (262.56) | 445.44 (577.53) | 867.78 (658.04)
  A/Wisconsin [CD4-IFNγ] | 492.75 (320.15) | 476.37 (416.85) | 548.14 (557.60) | 372.77 (618.70) | 399.91 (481.00) | 325.70 (547.57) | 523.69 (683.65) | 374.66 (407.51) | 467.74 (807.28) | 971.26 (783.42)
  B/Malaysia [CD4-IFNγ] | 522.75 (3348.47) | 510.43 (462.45) | 457.89 (774.10) | 253.06 (234.64) | 411.84 (384.77) | 240.48 (567.12) | 361.94 (357.95) | 360.90 (250.90) | 458.80 (456.80) | 1073.05 (935.35)
  A/Solomon Islands [CD4-IL2] | 316.88 (297.00) | 314.96 (372.22) | 558.83 (549.83) | 304.00 (404.11) | 368.31 (348.92) | 400.05 (505.26) | 304.33 (467.47) | 175.36 (258.68) | 691.47 (597.60) | 859.06 (642.57)
  A/Wisconsin [CD4-IL2] | 579.40 (330.85) | 426.54 (422.19) | 529.59 (677.44) | 480.46 (667.59) | 603.02 (608.61) | 551.29 (712.29) | 489.69 (841.98) | 339.94 (440.33) | 700.87 (861.25) | 1011.95 (565.94)
  B/Malaysia [CD4-IL2] | 549.00 (2767.21) | 617.40 (602.01) | 698.16 (823.21) | 315.90 (393.50) | 672.69 (432.34) | 373.28 (680.43) | 518.17 (374.93) | 345.05 (300.46) | 612.61 (455.63) | 1119.01 (801.11)
  A/Solomon Islands [CD4-TNFα] | 280.19 (284.35) | 188.48 (325.58) | 382.50 (490.32) | 200.30 (422.18) | 263.40 (301.07) | 350.38 (473.03) | 254.19 (373.61) | 228.89 (247.41) | 533.13 (517.19) | 730.49 (549.49)
  A/Wisconsin [CD4-TNFα] | 722.29 (288.16) | 600.27 (472.44) | 626.23 (655.14) | 395.86 (758.84) | 599.10 (496.66) | 512.38 (740.10) | 601.79 (703.08) | 561.14 (451.82) | 521.03 (873.58) | 1187.70 (734.12)
  B/Malaysia [CD4-TNFα] | 538.21 (2445.31) | 576.09 (352.91) | 408.52 (712.70) | 149.41 (359.72) | 476.90 (332.91) | 160.26 (542.67) | 360.57 (367.88) | 385.22 (227.19) | 505.39 (393.49) | 798.97 (716.33)

12. Secondary Outcome: The GM Number of Influenza-specific CD8 T-cells Per Million CD8+ T-cells for Each Vaccine Strain Producing at Least Two Different Immune Markers or Producing Each of the Immune Markers Plus Another Immune Marker at Days 0 and 21
Description: The markers assessed were Cluster of Differentiation 8-All doubles i.e. CD8-All doubles, CD8-CD40L, CD8-IFNγ, CD8-IL2 and CD8-TNFα. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Days 0 and 21
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD8 T-cells
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 24 | 19 | 25 | 24 | 24 | 23 | 23 | 23 | 23 | 23
cells per million CD8 T-cells
  A/Solomon Islands [CD8-All doubles] at Day 0 | 8.10 (135.40) | 12.90 (151.71) | 14.46 (122.65) | 3.25 (53.78) | 3.31 (91.60) | 2.31 (47.88) | 2.63 (98.13) | 6.83 (67.42) | 13.81 (116.94) | 7.69 (91.40)
  A/Solomon Islands [CD8-All doubles] at Day 21 | 7.45 (97.10) | 12.20 (127.89) | 9.54 (116.11) | 5.14 (87.63) | 4.87 (92.78) | 4.71 (49.37) | 9.62 (50.39) | 4.76 (132.76) | 6.33 (91.54) | 2.34 (132.36)
  A/Wisconsin [CD8-All doubles] at Day 0 | 9.69 (178.06) | 6.81 (126.03) | 9.85 (344.91) | 3.93 (124.78) | 6.67 (112.61) | 5.53 (169.17) | 8.19 (95.91) | 6.73 (108.10) | 8.22 (153.57) | 9.16 (63.84)
  A/Wisconsin [CD8-All doubles] at Day 21 | 31.08 (84.59) | 7.54 (234.23) | 9.77 (292.05) | 4.15 (66.82) | 7.73 (139.86) | 12.49 (189.06) | 16.86 (219.38) | 4.99 (168.28) | 39.03 (123.00) | 2.00 (57.24)
  B/Malaysia [CD8-All doubles] at Day 0 | 11.62 (200.31) | 15.68 (423.52) | 30.58 (282.37) | 10.85 (215.20) | 6.74 (63.87) | 2.48 (44.95) | 26.27 (218.28) | 23.57 (184.06) | 16.83 (232.88) | 11.02 (175.35)
  B/Malaysia [CD8-All doubles] at Day 21 | 42.50 (296.07) | 44.96 (351.05) | 20.54 (188.50) | 8.09 (302.34) | 31.02 (243.07) | 22.20 (183.56) | 60.96 (415.86) | 13.39 (193.75) | 24.91 (153.61) | 16.20 (225.18)
  A/Solomon Islands [CD8-CD40L] at Day 0 | 7.68 (76.49) | 9.18 (141.09) | 7.64 (81.73) | 2.31 (25.28) | 2.75 (106.31) | 1.47 (26.08) | 2.39 (55.56) | 2.94 (67.71) | 10.48 (95.48) | 2.70 (77.94)
  A/Solomon Islands [CD8-CD40L] at Day 21 | 3.76 (69.81) | 3.41 (98.02) | 8.71 (75.81) | 2.20 (47.58) | 3.22 (72.42) | 2.21 (42.86) | 3.36 (55.81) | 3.45 (82.08) | 2.30 (53.40) | 2.97 (43.37)
  A/Wisconsin [CD8-CD40L] at Day 0 | 4.63 (51.86) | 2.17 (41.97) | 5.20 (70.37) | 1.82 (70.40) | 2.78 (66.95) | 1.47 (26.82) | 3.10 (43.93) | 2.08 (53.94) | 4.55 (93.16) | 2.96 (99.03)
  A/Wisconsin [CD8-CD40L] at Day 21 | 3.09 (45.67) | 5.72 (165.77) | 4.19 (52.99) | 3.00 (45.24) | 5.72 (90.85) | 5.01 (88.79) | 5.58 (98.17) | 5.17 (34.65) | 7.27 (43.58) | 2.04 (35.04)
  B/Malaysia [CD8-CD40L] at Day 0 | 3.24 (54.73) | 7.16 (290.97) | 6.53 (132.89) | 2.82 (87.95) | 2.84 (47.37) | 1.66 (34.20) | 3.29 (76.69) | 5.21 (59.00) | 5.52 (168.72) | 3.98 (95.04)
  B/Malaysia [CD8-CD40L] at Day 21 | 2.68 (127.60) | 12.06 (265.01) | 3.74 (115.89) | 4.45 (142.55) | 9.13 (183.09) | 5.64 (138.31) | 8.97 (271.08) | 4.47 (183.70) | 3.43 (72.64) | 9.50 (127.97)
  A/Solomon Islands [CD8-IFNγ] at Day 0 | 7.38 (115.60) | 8.63 (157.70) | 10.16 (107.21) | 3.99 (62.89) | 4.69 (90.75) | 1.89 (57.50) | 3.04 (89.37) | 6.83 (63.62) | 8.68 (98.54) | 4.59 (65.86)
  A/Solomon Islands [CD8-IFNγ] at Day 21 | 7.37 (84.04) | 9.19 (85.93) | 11.15 (94.57) | 2.18 (51.19) | 3.96 (75.52) | 2.03 (23.00) | 5.60 (50.57) | 3.18 (106.55) | 3.25 (64.56) | 1.59 (141.41)
  A/Wisconsin [CD8-IFNγ] at Day 0 | 7.85 (103.62) | 3.95 (78.12) | 7.61 (309.89) | 2.46 (120.14) | 5.23 (75.71) | 2.51 (168.10) | 4.70 (53.61) | 4.05 (52.57) | 7.23 (129.33) | 7.26 (64.60)
  A/Wisconsin [CD8-IFNγ] at Day 21 | 8.27 (78.96) | 8.63 (176.22) | 9.89 (295.99) | 3.52 (66.86) | 6.18 (125.90) | 10.28 (119.10) | 12.07 (140.10) | 4.02 (92.71) | 6.94 (109.72) | 2.21 (47.90)
  B/Malaysia [CD8-IFNγ] at Day 0 | 5.56 (99.28) | 10.71 (390.44) | 15.15 (261.46) | 6.09 (157.93) | 10.28 (61.17) | 1.69 (19.96) | 17.27 (129.27) | 17.76 (137.26) | 9.94 (190.65) | 9.07 (168.50)
  B/Malaysia [CD8-IFNγ] at Day 21 | 11.69 (129.41) | 17.80 (305.22) | 14.44 (160.52) | 5.42 (269.73) | 14.05 (224.41) | 9.75 (159.06) | 23.95 (323.71) | 18.53 (162.45) | 21.99 (122.96) | 12.44 (163.33)
  A/Solomon Islands [CD8-IL2] at Day 0 | 3.52 (80.50) | 3.10 (27.39) | 5.50 (55.47) | 3.03 (42.10) | 1.20 (13.14) | 2.12 (30.13) | 3.28 (81.61) | 2.96 (40.40) | 4.00 (42.26) | 2.67 (38.98)
  A/Solomon Islands [CD8-IL2] at Day 21 | 4.80 (63.95) | 4.30 (73.39) | 7.50 (51.96) | 3.97 (61.17) | 1.98 (40.41) | 4.86 (57.41) | 4.36 (36.32) | 5.57 (83.12) | 7.30 (69.21) | 2.17 (44.90)
  A/Wisconsin [CD8-IL2] at Day 0 | 3.70 (113.92) | 3.21 (91.01) | 6.13 (99.85) | 3.13 (61.75) | 2.11 (71.74) | 4.05 (62.37) | 5.41 (65.29) | 6.43 (82.32) | 3.75 (71.92) | 2.00 (23.96)
  A/Wisconsin [CD8-IL2] at Day 21 | 12.45 (89.54) | 5.93 (78.91) | 7.70 (64.46) | 3.05 (40.35) | 2.97 (61.70) | 4.41 (109.49) | 10.92 (109.83) | 6.18 (125.87) | 14.11 (81.52) | 2.69 (51.22)
  B/Malaysia [CD8-IL2] at Day 0 | 8.66 (147.36) | 4.40 (161.85) | 10.05 (141.49) | 9.50 (106.18) | 2.13 (22.15) | 2.66 (49.28) | 12.10 (182.42) | 17.14 (88.20) | 6.41 (108.44) | 2.17 (64.13)
  B/Malaysia [CD8-IL2] at Day 21 | 17.85 (257.14) | 32.92 (72.84) | 9.72 (118.83) | 4.83 (129.69) | 7.60 (27.90) | 8.49 (137.21) | 17.98 (127.27) | 5.19 (81.07) | 7.95 (75.16) | 12.46 (96.16)
  A/Solomon Islands [CD8-TNFα] at Day 0 | 5.41 (91.54) | 3.26 (34.12) | 8.71 (71.14) | 2.59 (42.20) | 2.58 (39.14) | 2.28 (45.26) | 2.18 (33.72) | 5.63 (58.18) | 3.94 (52.44) | 4.33 (81.83)
  A/Solomon Islands [CD8-TNFα] at Day 21 | 3.79 (79.93) | 12.15 (70.97) | 2.76 (117.87) | 5.85 (65.60) | 2.68 (61.45) | 3.78 (51.36) | 5.33 (36.95) | 6.03 (110.26) | 4.35 (64.50) | 1.91 (131.67)
  A/Wisconsin [CD8-TNFα] at Day 0 | 5.04 (145.40) | 3.70 (138.04) | 5.31 (338.73) | 3.70 (67.70) | 8.64 (86.13) | 9.54 (187.33) | 5.96 (128.54) | 10.06 (78.63) | 3.93 (93.43) | 3.41 (64.37)
  A/Wisconsin [CD8-TNFα] at Day 21 | 14.64 (98.80) | 5.75 (118.21) | 5.74 (278.42) | 3.47 (65.17) | 5.60 (66.01) | 12.32 (188.66) | 11.29 (211.80) | 8.52 (135.47) | 16.28 (142.20) | 2.52 (46.95)
  B/Malaysia [CD8-TNFα] at Day 0 | 11.49 (167.40) | 11.28 (215.17) | 18.47 (194.16) | 8.77 (177.85) | 6.77 (50.82) | 2.67 (37.22) | 26.25 (172.19) | 23.27 (109.52) | 14.97 (169.37) | 9.07 (123.64)
  B/Malaysia [CD8-TNFα] at Day 21 | 28.50 (261.61) | 13.76 (122.97) | 9.28 (142.76) | 9.21 (224.57) | 15.20 (160.37) | 9.02 (96.93) | 27.84 (355.89) | 15.64 (126.07) | 19.42 (124.13) | 8.57 (151.66)

13. Secondary Outcome: The GM Number of Influenza-specific CD8 T-cells Per Million CD8+ T-cells for Each Vaccine Strain Producing at Least Two Different Immune Markers or Producing Each of the Immune Markers Plus Another Immune Marker at Day 180
Description: The markers assessed were CD8-All doubles, CD8-CD40L, CD8-IFNγ, CD8-IL2 and CD8-TNFα. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 180
Population: Analysis was performed on According-to-Protocol (ATP) cohort for persistence for cell mediated immunity (CMI) which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available at day 180.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD8 T-cells
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 21 | 18 | 20 | 17 | 21 | 20 | 19 | 16 | 16 | 19
cells per million CD8 T-cells
  A/Solomon Islands [CD8-All doubles] | 2.57 (89.78) | 14.64 (96.62) | 3.61 (143.10) | 4.75 (74.09) | 3.05 (107.06) | 1.24 (15.43) | 2.64 (47.18) | 4.81 (90.76) | 7.32 (115.74) | 5.64 (98.76)
  A/Wisconsin [CD8-All doubles] | 21.14 (506.65) | 9.63 (110.40) | 18.10 (367.31) | 16.14 (132.83) | 20.72 (412.35) | 21.73 (368.70) | 21.00 (327.24) | 11.95 (384.28) | 10.44 (226.57) | 3.13 (186.12)
  B/Malaysia [CD8-All doubles] | 9.92 (111.75) | 7.10 (132.35) | 12.14 (319.23) | 9.61 (157.68) | 25.48 (138.45) | 9.18 (143.21) | 12.73 (460.97) | 4.71 (115.31) | 6.47 (83.62) | 7.96 (132.07)
  A/Solomon Islands [CD8-CD40L] | 2.92 (53.08) | 12.64 (119.84) | 2.95 (97.98) | 3.18 (74.24) | 3.97 (69.10) | 1.93 (31.31) | 2.70 (59.56) | 4.89 (86.67) | 8.74 (100.11) | 3.94 (40.79)
  A/Wisconsin [CD8-CD40L] | 18.75 (312.61) | 7.79 (60.25) | 10.73 (230.49) | 15.32 (145.70) | 9.60 (232.78) | 8.57 (321.14) | 13.90 (118.80) | 6.00 (315.87) | 6.46 (135.88) | 3.43 (66.51)
  B/Malaysia [CD8-CD40L] | 5.79 (103.71) | 5.64 (75.90) | 10.61 (125.46) | 7.48 (92.38) | 8.46 (105.02) | 6.10 (113.43) | 3.77 (59.02) | 2.75 (73.05) | 3.63 (81.37) | 3.78 (95.38)
  A/Solomon Islands [CD8-IFNγ] | 2.00 (54.66) | 3.12 (124.76) | 3.13 (50.16) | 3.89 (53.23) | 1.90 (35.38) | 3.12 (47.02) | 3.07 (31.51) | 3.11 (45.39) | 2.36 (55.08) | 2.65 (79.58)
  A/Wisconsin [CD8-IFNγ] | 4.21 (167.18) | 2.68 (42.60) | 2.32 (92.50) | 2.89 (43.98) | 2.50 (53.46) | 2.53 (46.46) | 2.39 (154.17) | 3.67 (78.90) | 1.97 (157.41) | 2.72 (125.70)
  B/Malaysia [CD8-IFNγ] | 10.63 (76.06) | 3.72 (66.40) | 6.46 (183.07) | 6.19 (170.54) | 10.24 (49.87) | 4.96 (55.70) | 8.54 (430.43) | 2.56 (40.61) | 4.12 (49.87) | 5.33 (182.33)
  A/Solomon Islands [CD8-IL2] | 1.97 (64.78) | 10.49 (74.37) | 2.82 (105.05) | 3.36 (44.53) | 3.76 (68.56) | 1.89 (25.49) | 4.31 (70.92) | 4.89 (86.67) | 4.93 (111.36) | 7.15 (75.19)
  A/Wisconsin [CD8-IL2] | 20.60 (427.25) | 15.24 (108.11) | 14.05 (351.12) | 42.75 (112.35) | 19.37 (415.28) | 32.48 (357.67) | 15.96 (296.44) | 11.89 (385.26) | 10.37 (212.91) | 4.04 (153.21)
  B/Malaysia [CD8-IL2] | 4.15 (92.98) | 7.59 (100.66) | 11.05 (217.46) | 7.47 (77.13) | 11.50 (130.60) | 11.62 (176.05) | 3.86 (81.13) | 5.99 (110.92) | 4.38 (95.85) | 6.11 (91.97)
  A/Solomon Islands [CD8-TNFα] | 2.54 (60.55) | 2.35 (31.14) | 2.09 (62.82) | 3.60 (37.07) | 1.62 (76.42) | 1.53 (21.24) | 2.44 (28.80) | 2.73 (44.50) | 2.54 (79.84) | 3.39 (69.30)
  A/Wisconsin [CD8-TNFα] | 7.78 (244.26) | 4.42 (63.49) | 9.25 (151.69) | 6.69 (85.85) | 6.67 (210.64) | 3.26 (108.02) | 9.09 (213.44) | 4.86 (78.63) | 6.81 (139.38) | 3.52 (125.46)
  B/Malaysia [CD8-TNFα] | 4.05 (74.16) | 5.66 (88.74) | 14.08 (191.59) | 3.84 (93.04) | 6.11 (48.41) | 5.46 (88.95) | 5.07 (415.90) | 3.63 (81.27) | 4.69 (42.36) | 4.58 (132.21)

14. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 ecchymosis, pain, redness and swelling was greater than 100 millimeter (mm) i.e. > 100 mm and grade 3 pain was considerable pain at rest that prevented normal everyday activities. Any was occurrence of any local symptom regardless of their intensity grade. Any for ecchymosis, redness and swelling was >20mm.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 201 | 201 | 201 | 201 | 198 | 197 | 198 | 198 | 200 | 201
Subjects
  Any ecchymosis | 3 | 1 | 5 | 1 | 2 | 2 | 4 | 2 | 3 | 0
  Grade 3 ecchymosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any pain | 68 | 82 | 111 | 84 | 91 | 119 | 93 | 106 | 32 | 93
  Grade 3 pain | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
  Any redness | 15 | 16 | 37 | 12 | 33 | 36 | 18 | 34 | 5 | 2
  Grade 3 redness | 0 | 1 | 3 | 1 | 1 | 2 | 0 | 2 | 0 | 0
  Any swelling | 13 | 12 | 25 | 13 | 18 | 23 | 11 | 25 | 5 | 2
  Grade 3 swelling | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0

15. Secondary Outcome: Duration of Solicited Local AEs
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom and completed information on duration in their symptom sheet.
Measure: Median (Full Range); unit: Days
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 68 | 82 | 111 | 84 | 91 | 119 | 93 | 106 | 32 | 93
Days
  Ecchymosis (N=3;1;5;1;2;2;4;2;3;0) | 5.0 [1.0 to 7.0] | 6.0 [6.0 to 6.0] | 6.0 [3.0 to 7.0] | 2.0 [2.0 to 2.0] | 2.5 [1.0 to 4.0] | 3.0 [1.0 to 5.0] | 3.0 [1.0 to 5.0] | 3.0 [2.0 to 4.0] | 5.0 [4.0 to 7.0] | NA [NA to NA] — None of the subjects in this group reported any ecchymosis.
  Pain (N=68;82;111;84;91;119;93;106;32;93) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Redness (N=14;16;35;11;33;36;18;34;5;2) | 1.5 [1.0 to 5.0] | 2.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0] | 3.0 [1.0 to 6.0] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0]
  Swelling (N=12;12;24;12;17;23;11;25;5;2) | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 6.0] | 2.5 [1.0 to 7.0] | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0] | 1.5 [1.0 to 2.0]

16. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any Fever was defined as axillary temperature greater than or equal to 38.0 degree centigrade i.e.≥ 38.0°C, grade 3 fever was axillary temperature >40°C. For other symptoms, any was defined as occurrence of any general symptom regardless of intensity grade or relation to vaccination and grade 3 was defined as a general symptom that prevented normal activity. Related was a general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 201 | 201 | 201 | 201 | 198 | 198 | 198 | 198 | 200 | 201
Subjects
  Any arthralgia | 15 | 23 | 36 | 16 | 21 | 45 | 28 | 35 | 16 | 12
  Grade 3 arthralgia | 3 | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 0
  Related arthralgia | 11 | 15 | 30 | 10 | 16 | 28 | 20 | 25 | 9 | 9
  Any fatigue | 34 | 35 | 54 | 35 | 46 | 55 | 38 | 63 | 24 | 41
  Grade 3 fatigue | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Related fatigue | 21 | 24 | 39 | 20 | 35 | 38 | 25 | 35 | 16 | 30
  Any headache | 22 | 38 | 47 | 35 | 39 | 55 | 36 | 48 | 23 | 45
  Grade 3 headache | 2 | 1 | 2 | 0 | 0 | 4 | 0 | 1 | 0 | 0
  Related headache | 14 | 23 | 28 | 18 | 24 | 27 | 15 | 27 | 20 | 30
  Any myalgia | 20 | 35 | 57 | 30 | 47 | 66 | 46 | 56 | 19 | 40
  Grade 3 myalgia | 1 | 1 | 2 | 1 | 1 | 3 | 0 | 2 | 0 | 1
  Related myalgia | 13 | 29 | 46 | 24 | 36 | 46 | 34 | 44 | 15 | 33
  Any nausea | 10 | 12 | 19 | 10 | 13 | 18 | 8 | 14 | 6 | 13
  Grade 3 nausea | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Related nausea | 6 | 9 | 10 | 5 | 8 | 9 | 4 | 10 | 4 | 11
  Any shivering | 13 | 18 | 37 | 26 | 18 | 43 | 17 | 31 | 8 | 21
  Grade 3 shivering | 1 | 3 | 2 | 0 | 0 | 4 | 0 | 2 | 0 | 1
  Related shivering | 9 | 14 | 26 | 21 | 7 | 27 | 12 | 21 | 6 | 16
  Any fever | 1 | 1 | 3 | 2 | 2 | 6 | 3 | 6 | 0 | 1
  Grade 3 fever | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related fever | 1 | 1 | 3 | 2 | 1 | 5 | 3 | 4 | 0 | 1

17. Secondary Outcome: Duration of Solicited General AEs
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: as for outcome 15
Measure: Median (Full Range); unit: Days
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 34 | 38 | 57 | 35 | 47 | 66 | 46 | 63 | 24 | 45
Days
  Arthralgia (N=15;23;36;16;21;45;28;35;16;12) | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Fatigue (N=34;35;54;35;46;55;38;63;24;41) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Headache (N=22;38;47;35;39;55;36;48;23;45) | 1.5 [1.0 to 7.0] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 5.0] | 1.5 [1.0 to 6.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0]
  Myalgia (N=20;35;57;30;47;66;46;56;19;40) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Nausea (N=10;12;19;10;13;18;8;14;6;13) | 1.5 [1.0 to 4.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 5.0] | 1.5 [1.0 to 5.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 7.0] | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 6.0]
  Shivering (N=13;18;37;26;18;43;17;31;8;21) | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0] | 2.5 [1.0 to 7.0] | 1.0 [1.0 to 6.0]
  Fever (N=4;3;9;4;3;14;6;12;0;1) | 1.0 [1.0 to 1.0] | 3.0 [3.0 to 3.0] | 1.5 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | NA [NA to NA] — None of the subjects in this group reported any fever. | 1.0 [1.0 to 1.0]

18. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During a 21-day follow-up period (Day 0-20) after vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 204 | 202 | 202 | 202 | 199 | 198 | 198 | 199 | 200 | 203
Subjects
  Any AE(s) | 41 | 32 | 51 | 39 | 34 | 42 | 34 | 43 | 27 | 44
  Grade 3 AE(s) | 1 | 3 | 8 | 3 | 0 | 6 | 1 | 6 | 1 | 3
  Related AE(s) | 5 | 7 | 15 | 6 | 13 | 13 | 8 | 18 | 6 | 13

19. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Adverse Events Resulting in Medically Attended Visit Between Day 0 and Day 20
Description: For each solicited and unsolicited AE the subject experienced, the subject was asked if they had received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and grade 3 was defined as a symptom that prevented normal activity. Related was a symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Between Day 0 and Day 20 after vaccination
Population: as for outcome 18
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 204 | 202 | 202 | 202 | 199 | 198 | 198 | 199 | 200 | 203
Subjects
  Any AE(S) | 15 | 10 | 19 | 15 | 16 | 14 | 11 | 13 | 10 | 13
  Grade 3 AE(s) | 0 | 2 | 4 | 3 | 0 | 4 | 1 | 4 | 1 | 1
  Related AE(s) | 0 | 0 | 4 | 0 | 1 | 2 | 0 | 2 | 1 | 2

20. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Adverse Events Resulting in Medically Attended Visit Between Day 21 and Day 179
Description: as for outcome 19
Time Frame: Between Day 21 and Day 179 after vaccination
Population: as for outcome 18
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 204 | 202 | 202 | 202 | 199 | 198 | 198 | 199 | 200 | 203
Subjects
  Any AE (s) | 78 | 60 | 79 | 71 | 65 | 67 | 67 | 69 | 69 | 62
  Grade 3 AE(s) | 18 | 11 | 13 | 13 | 10 | 12 | 17 | 15 | 17 | 10
  Related AE(s) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

21. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) Between Day 0 and Day 20
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Between Day 0 and Day 20 after vaccination
Population: as for outcome 18
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 204 | 202 | 202 | 202 | 199 | 198 | 198 | 199 | 200 | 203
Subjects
  Any SAE(s) | 0 | 3 | 2 | 2 | 2 | 4 | 2 | 4 | 0 | 0
  Related SAE(s) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

22. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) Between Day 21 and Day 179
Description: as for outcome 21
Time Frame: Between Day 21 and Day 179 after vaccination
Population: as for outcome 18
Measure: Number; unit: Subjects
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 204 | 202 | 202 | 202 | 199 | 198 | 198 | 199 | 200 | 203
Subjects
  Any SAE(s) | 18 | 9 | 5 | 8 | 9 | 10 | 16 | 19 | 15 | 3
  Related SAE(s) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from day 0 to day 20 and day 21 to day 179. Systematically assessed frequent adverse events (AEs) and non-systematically assessed frequent AEs were assessed during 7 day and 21 day post vaccination period respectively.
Description: For the systematically assessed other (non-serious) adverse events,the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | Influenza Vaccine GSK576389A Formulation 1 Group | Influenza Vaccine GSK576389A Formulation 2 Group | Influenza Vaccine GSK576389A Formulation 3 Group | Influenza Vaccine GSK576389A Formulation 4 Group | Influenza Vaccine GSK576389A Formulation 5 Group | Influenza Vaccine GSK576389A Formulation 6 Group | Influenza Vaccine GSK576389A Formulation 7 Group | Influenza Vaccine GSK576389A Formulation 8 Group | Fluarix Elderly Group | Fluarix Young Group
Serious Adverse Events (participants affected / at risk) | 18/204 | 9/202 | 5/202 | 8/202 | 9/199 | 10/198 | 16/198 | 19/199 | 15/200 | 3/203
Other Adverse Events (participants affected / at risk) | 107/204 | 129/202 | 150/202 | 121/202 | 138/199 | 158/198 | 134/198 | 155/199 | 74/200 | 133/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine GSK576389A Formulation 1 Group (N=204) | Influenza Vaccine GSK576389A Formulation 2 Group (N=202) | Influenza Vaccine GSK576389A Formulation 3 Group (N=202) | Influenza Vaccine GSK576389A Formulation 4 Group (N=202) | Influenza Vaccine GSK576389A Formulation 5 Group (N=199) | Influenza Vaccine GSK576389A Formulation 6 Group (N=198) | Influenza Vaccine GSK576389A Formulation 7 Group (N=198) | Influenza Vaccine GSK576389A Formulation 8 Group (N=199) | Fluarix Elderly Group (N=200) | Fluarix Young Group (N=203)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 — Assessed between Day 0 and Day 20
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 0 and Day 20
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 0 and Day 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 0 and Day 20
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 0 and Day 20
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 0 and Day 20
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 0 and Day 20
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Assessed between Day 0 and Day 20
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 0 and Day 20
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 — Assessed between Day 21 and Day 179
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 — Assessed between Day 21 and Day 179
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 — Assessed between Day 21 and Day 179
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Bifascicular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Assessed between Day 21 and Day 179
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Assessed between Day 21 and Day 179
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Assessed between Day 21 and Day 179
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Assessed between Day 21 and Day 179
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Assessed between Day 21 and Day 179
Vestibular neuronitis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Assessed between Day 21 and Day 179
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Influenza Vaccine GSK576389A Formulation 1 Group (N=204) | Influenza Vaccine GSK576389A Formulation 2 Group (N=202) | Influenza Vaccine GSK576389A Formulation 3 Group (N=202) | Influenza Vaccine GSK576389A Formulation 4 Group (N=202) | Influenza Vaccine GSK576389A Formulation 5 Group (N=199) | Influenza Vaccine GSK576389A Formulation 6 Group (N=198) | Influenza Vaccine GSK576389A Formulation 7 Group (N=198) | Influenza Vaccine GSK576389A Formulation 8 Group (N=199) | Fluarix Elderly Group (N=200) | Fluarix Young Group (N=203)
Pain (General disorders) | 68/201 | 82/201 | 111/201 | 84/201 | 91/198 | 119/197 | 93 | 106/198 | 32 | 93/201
Redness (General disorders) | 15/201 | 16/201 | 37/201 | 12/201 | 33/198 | 36/197 | 18 | 34/198 | 5 | 2/201
Swelling (General disorders) | 13/201 | 12/201 | 25/201 | 13/201 | 18/198 | 23/197 | 11 | 25/198 | 5 | 2/201
Arthralgia (General disorders) | 15/201 | 23/201 | 36/201 | 16/201 | 21/198 | 45 | 28 | 35/198 | 16 | 12/201
Fatigue (General disorders) | 34/201 | 35/201 | 54/201 | 35/201 | 46/198 | 55 | 38 | 63/198 | 24 | 41/201
Headache (General disorders) | 22/201 | 38/201 | 47/201 | 35/201 | 39/198 | 55 | 36 | 48/198 | 23 | 45/201
Myalgia (General disorders) | 20/201 | 35/201 | 57/201 | 30/201 | 47/198 | 66 | 46 | 56/198 | 19 | 40/201
Nausea (General disorders) | 10/201 | 12/201 | 19/201 | 10/201 | 13/198 | 18 | 8 | 14/198 | 6 | 13/201
Shivering (General disorders) | 13/201 | 18/201 | 37/201 | 26/201 | 18/198 | 43 | 17 | 31/198 | 8 | 21/201
Nasopharyngitis (Infections and infestations) | 9 | 4 | 7 | 5 | 7 | 8 | 6 | 7 | 2 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.